CLINICAL TRIAL: NCT04866069
Title: Phase I Study Evaluating the Safety and Efficacy of the Protective Adjuvanted Inactivated Vaccine Developed Against SARS-CoV-2 in Healthy Participants, Administered as Two Injections Subcutaneously in Two Different Dosages.
Brief Title: Study of a Severe Acute Respiratory Syndrome-Coronavirus-2 (SARS-CoV-2) Adjuvanted Inactivated Vaccine in Healthy Adults
Acronym: COVID-19
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Although cellular responses to virus were satisfactory, neutralizing titres against virus were lower then expected levels
Sponsor: Osman ERGANIS, PhD, Prof (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other); VETAL Inc. (Unknown); MonitorCRO (Industry)
Responsible Party: Sponsor-Investigator, Osman ERGANIS, PhD, Prof, PhD, Prof, The Scientific and Technological Research Council of Turkey
Organization: The Scientific and Technological Research Council of Turkey (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ISV2AOH3ODN
Record Dates: First submitted 2021-04-26; First posted 2021-04-29 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Covid19
Keywords: SARS-CoV-2; Adjuvanted inactivated vaccine
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low-Dose Group (Group A) (Experimental): 20 participants will receive 10 µg-3M inactivated virus + 1 mg Al(OH)3 + 300 µg CpGODN adjuvanted vaccine
  Interventions: Biological: SARS-CoV-2 vaccine
- High-Dose Group (Group B) (Experimental): 20 participants will receive 20 µg-6M inactivated virus + 1 mg Al(OH)3 + 300 µg CpGODN adjuvanted vaccine
  Interventions: Biological: SARS-CoV-2 vaccine
- Placebo Group (Placebo Comparator): 10 participants will receive 1 ml of 0.9% sodium chloride (NaCl)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: SARS-CoV-2 vaccine — Adjuvanted inactivated vaccine
  Arms: High-Dose Group (Group B); Low-Dose Group (Group A)
Biological: Placebo — 0.9% NaCl
  Arms: Placebo Group

SUMMARY:
This phase I study is designed as double-blinded, randomised, placebo controlled, three-armed study composed of two different dose arms of protective adjuvanted inactivated vaccine against SARS-CoV-2 in dose escalations (first low dose group, followed by high dose group) and placebo arm.

DETAILED DESCRIPTION:
This phase I study is designed as double-blinded, randomised, placebo controlled, three-armed study composed of two different dose arms of protective adjuvanted inactivated vaccine against SARS-CoV-2 in dose escalations (first low dose group, followed by high dose group) and placebo arm. Each dose of vaccine will be defined as a cohort in itself, with vaccine administration to 20 participants and placebo administration to 5 participants. After completion of low-dose group, decision of switch to high-dose will be taken by the Independent Data Monitoring Committee and will continue accordingly.

In the study, 50 healthy participants of 18-45 years of age will be recruited.

All injections will be done subcutaneously.

Injections will be administered at 1 and 21 days.

The participants will be followed for 6 months and the study will be completed in 12 months.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for the study, each participant must satisfy all the following criteria:

1. Healthy participants between 18-45 years of age,
2. Sign an informed consent document,
3. Negative immunoglobulin G (IgG) and immunoglobulin M (IgM) antibody for COVID-19,
4. Negative quantitative polymerase chain reaction (qPCR) SARS-CoV-2 results of nasopharyngeal/sputum samples,
5. Able to comply with the study protocol during the study period,
6. Negative tests for Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV), Hepatitis C Virus (HCV),
7. Body temperature <37.2 C and no signs of active infection,
8. Body mass index 18-35 kg/m2,
9. Normal laboratory levels of whole blood count, alanine transaminase (ALT), aspartate transaminase (AST), total bilirubin, urea, creatinine, and fasting blood glucose, or abnormal finding detected in any laboratory parameter which is not greater than Grade 1 according to the investigator's evaluation,
10. Good general health (no known disease in the history and physical examination within 14 days prior to the enrolment),
11. Female and male participants who will be able to have appropriate contraception methods within 30 days prior to vaccine injection and within 6 months after vaccination,

Exclusion Criteria:

Participants with any of the following criteria will be excluded:

1. History of seizure, encephalopathy, or psychosis,
2. History of allergic reactions to any known vaccine or to any component of the study vaccine,
3. Pregnant, breastfeeding, or positive pregnancy test or planning to conceive within 6 months,
4. History of SARS-CoV-2 infection,
5. Severe cardiovascular disorders (arrhythmia, conduction disorders, history of myocardial infarction, uncontrolled hypertension),
6. Severe chronic disorders (asthma, diabetes mellitus, thyroid disorders…etc),
7. Congenital or acquired angioedema,
8. Diagnosis of immunodeficiency,
9. Diagnosis of bleeding diathesis,
10. Use of immunosuppressive treatment, anti-allergic treatment, cytotoxic treatment, inhaler corticosteroids (allergic rhinitis or topical steroid ointments are excluded),
11. Those who received blood and blood product transfusions in the last 6 months,
12. Those on any vaccine program or experimental medication within 1 month prior to the study,
13. History of any vaccination against SARS-CoV-2 within 1 month prior to the study,
14. Use of active tuberculosis treatment,
15. History of addictive drug use,
16. History of alcohol abuse and/or history of alcohol intake more than 2 units per day or 10 units per week and/or positive breath alcohol test (one unit of alcohol equals to 250 mL beer, 125 mL wine or 25 mL whiskey),
17. According to the investigator's evaluation, those who have any condition (medical, psychological, social, etc.) that may impair the patient's compliance with the study will be excluded from the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2021-04-25 (Actual); Primary Completion 2021-09-05 (Actual); Study Completion 2021-09-05 (Actual)

PRIMARY OUTCOMES:
Acute adverse events (AEs) | 24 hours
  Frequency of acute adverse events in all dosage groups
Solicited local and systemic adverse events (AEs) | 15 days
  Frequency of local and systemic AEs in all dosage groups
Unsolicited local and systemic adverse events (AEs) | 28 days
  Frequency of local and systemic AEs in all dosage groups

SECONDARY OUTCOMES:
Neutralizing antibody response | Before first dose administration, on Day 21-28-35 and Month 3 and Month 6 after first dose administration.
  Immunogenicity response by measuring neutralizing antibody titer (anti-spike and anti-RBD) developed against SARS-CoV-2 (by ELISA)
Cellular immune response | Before first dose administration, on Day 21-28-35 and Month 3 and Month 6 after first dose administration.
  Interferon-γ (IFN-γ) positive cell level (by ELISPOT)

CONTACTS AND LOCATIONS:
Overall Officials: Oguz Akbas, MD, Study Director — MonitorCRO
Locations (1):
- Ankara City Hospital Phase I Drug Research Center, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No